CLINICAL TRIAL: NCT06657911
Title: SUBLIME: Size Up Bicuspid with the LIra MEthod: the SUBLIME Study
Brief Title: Size Up Bicuspid with the LIra MEthod: the SUBLIME Study
Acronym: SUBLIME
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Matteo Montorfano, Professor, cardiologist, IRCCS San Raffaele
Other Study IDs: SUBLIME
Record Dates: First submitted 2024-09-24; First posted 2024-10-26 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Bicuspid Aortic Valve (BAV)
Keywords: LIRA method; Bicuspid aortic Valve; TAVR
MeSH Terms: conditions — Bicuspid Aortic Valve Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- BAV patients underoging TAVR: Patients with bicuspid aortic valve undergoing TAVI for severe aortic stenosis with sizing performed

SUMMARY:
Transcatheter aortic valve replacement (TAVR) outcomes in patients with raphe-type bicuspid aortic valve (BAV) are still suboptimal for the non negligible rate of stroke and permanent pacemaker implantation. There is still lack of consensus on the optimal sizing method for prosthesis selection in BAV patients.

The objective of the present study is to evaluate the efficacy and safety of the LIRA sizing method in raphe-type BAV patients undergoing TAVR.

DETAILED DESCRIPTION:
Bicuspid aortic valve (BAV) still represents a challenge for percutaneous treatment due to the peculiar anatomy.

BAV patients have been historically excluded from major randomized controlled trials.

Observational data have showed a high rate of paravalvular leak (PVL) with the use of self-expanding prostheses and a non-negligible rate of annular rupture with the use of balloon expandable valves.

More recent data have shown better outcomes with current generation prostheses although the rate of stroke and permanent pacemaker implantation remains high.

These suboptimal results, possibly related to BAV different anatomy, have advocated the use of different sizing method for prosthesis selection in this setting.

Recent evidence has shown that transcatheter heart valve (THV) anchoring in BAV patients might occur at the raphe-level, defined as the LIRA (Level of Implantation at the RAphe) plane. Thus, a novel supra-annular sizing method based on the measurement of the perimeter at the raphe-level, the LIRA-method, has been developed in our center and validated in small cohorts of patients.

The aim of our study is to evaluate the efficacy and safety of the LIRA method in raphe-type bicuspid patients undergoing TAVR.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years old with severe aortic stenosis and type 1 or 2 BAV according to Sievers classification) undergone TAVR with self-expanding supra-annular prostheses sized according to the LIRA method between September 2018 and June 2024

Exclusion Criteria:

* Redo-TAVR
* TAVR performed in emergency setting
* TAVR performed for severe aortic regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 18 years old with severe aortic stenosis and type 1 or 2 BAV undergone TAVR with self-expanding supra-annular prostheses sized according to the LIRA method
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-12-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Device success | Up to 30 days after TAVI procedure
  Device success as defined by VARC 3 criteria : presence of technical success, freedom from mortality, freedom from surgery or intervention related to the device or to a major vascular or access-related or cardiac structural complications, intended performance of the valve (less than moderate aortic regurgitation, mean gradient < 20 mmHg, peak velocity <3 m/s, doppler velocity index >0.25).

SECONDARY OUTCOMES:
Number of partecipants with TAVI-related Adverse Events as assessed by VARC 3 criteria. | Up to 30 days after TAVI procedure
  * All-cause mortality
  * All stroke
  * VARC type 2-4 bleeding
  * Major vascular, access-related, or cardiac structural complication
  * Acute kidney injury stage 3 or 4
  * New permanent pacemaker due to procedure- related conduction abnormalities
  * Surgery or intervention related to the device
Clinical efficacy | Up to 1 year after TAVI procedure
  Freedom from all-cause mortality, freedom from all stroke, freedom from hospitalization for procedure -or-valve-related causes, freedom from KCCQ Overall Summary score <45 or decline from baseline >10 point
Technical success | At exit from procedure room
  Freedom from mortality; successful access, delivery and retrieval of the delivery system; correct positioning of a single prosthetic heart valve into the proper anatomical location; freedom from surgey or intervention related to the device or to a major vascular or access-related, or cardiac structural.
Intended performance of the valve | Up to 30 days after TAVI procedure
  Less than moderate aortic regurgitation, mean gradient < 20 mmHg, peak velocity <3 m/s, doppler velocity index >0.25

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Matteo Montorfano, MD, Principal Investigator — IRCCS San Raffaele Scientific Institute
Locations (5):
- Italy (4):
  - Fondazione Poliambulanza, Brescia, Italy
  - Spedali Civili, Brescia, Italy
  - Ospedale San Donato, Milan, Italy
  - San Camillo Hospital, Roma, Italy
- Luzerner Kantonsspital, Lucerne, Switzerland, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hayashida K, Bouvier E, Lefevre T, Chevalier B, Hovasse T, Romano M, Garot P, Watanabe Y, Farge A, Donzeau-Gouge P, Cormier B, Morice MC. Transcatheter aortic valve implantation for patients with severe bicuspid aortic valve stenosis. Circ Cardiovasc Interv. 2013 Jun;6(3):284-91. doi: 10.1161/CIRCINTERVENTIONS.112.000084. Epub 2013 Jun 11. PMID 23756698
- [Background] Bauer T, Linke A, Sievert H, Kahlert P, Hambrecht R, Nickenig G, Hauptmann KE, Sack S, Gerckens U, Schneider S, Zeymer U, Zahn R. Comparison of the effectiveness of transcatheter aortic valve implantation in patients with stenotic bicuspid versus tricuspid aortic valves (from the German TAVI Registry). Am J Cardiol. 2014 Feb 1;113(3):518-21. doi: 10.1016/j.amjcard.2013.10.023. Epub 2013 Nov 9. PMID 24342758
- [Background] Perlman GY, Blanke P, Dvir D, Pache G, Modine T, Barbanti M, Holy EW, Treede H, Ruile P, Neumann FJ, Gandolfo C, Saia F, Tamburino C, Mak G, Thompson C, Wood D, Leipsic J, Webb JG. Bicuspid Aortic Valve Stenosis: Favorable Early Outcomes With a Next-Generation Transcatheter Heart Valve in a Multicenter Study. JACC Cardiovasc Interv. 2016 Apr 25;9(8):817-824. doi: 10.1016/j.jcin.2016.01.002. PMID 27101906
- [Background] Yoon SH, Lefevre T, Ahn JM, Perlman GY, Dvir D, Latib A, Barbanti M, Deuschl F, De Backer O, Blanke P, Modine T, Pache G, Neumann FJ, Ruile P, Arai T, Ohno Y, Kaneko H, Tay E, Schofer N, Holy EW, Luk NHV, Yong G, Lu Q, Kong WKF, Hon J, Kao HL, Lee M, Yin WH, Park DW, Kang SJ, Lee SW, Kim YH, Lee CW, Park SW, Kim HS, Butter C, Khalique OK, Schaefer U, Nietlispach F, Kodali SK, Leon MB, Ye J, Chevalier B, Leipsic J, Delgado V, Bax JJ, Tamburino C, Colombo A, Sondergaard L, Webb JG, Park SJ. Transcatheter Aortic Valve Replacement With Early- and New-Generation Devices in Bicuspid Aortic Valve Stenosis. J Am Coll Cardiol. 2016 Sep 13;68(11):1195-1205. doi: 10.1016/j.jacc.2016.06.041. PMID 27609682
- [Background] Iannopollo G, Romano V, Buzzatti N, De Backer O, Sondergaard L, Merkely B, Prendergast BD, Giannini F, Colombo A, Latib A, Granada JF, Chieffo A, Montorfano M. A novel supra-annular plane to predict TAVI prosthesis anchoring in raphe-type bicuspid aortic valve disease: the LIRA plane. EuroIntervention. 2020 Jun 25;16(3):259-261. doi: 10.4244/EIJ-D-19-00951. No abstract available. PMID 31659989
- [Background] Iannopollo G, Romano V, Buzzatti N, Ancona M, Ferri L, Russo F, Bellini B, Granada JF, Chieffo A, Montorfano M. Supra-annular sizing of transcatheter aortic valve prostheses in raphe-type bicuspid aortic valve disease: the LIRA method. Int J Cardiol. 2020 Oct 15;317:144-151. doi: 10.1016/j.ijcard.2020.05.076. Epub 2020 May 28. PMID 32473284
- [Background] Iannopollo G, Romano V, Esposito A, Guazzoni G, Ancona M, Ferri L, Russo F, Bellini B, Buzzatti N, Curio J, Prendergast B, Montorfano M. Update on supra-annular sizing of transcatheter aortic valve prostheses in raphe-type bicuspid aortic valve disease according to the LIRA method. Eur Heart J Suppl. 2022 May 18;24(Suppl C):C233-C242. doi: 10.1093/eurheartj/suac014. eCollection 2022 May. PMID 35602251